CLINICAL TRIAL: NCT03617757
Title: Determinants of Progression From Impaired Fasting Glucose to Diabetes Mellitus Among Chinese - a 3-year Follow up Study
Brief Title: Progression From Impaired Fasting Glucose to Diabetes Mellitus Among Chinese
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. YU Yee Yak, Esther, Clinical Assistant Professor, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: UW17-429
Record Dates: First submitted 2018-06-26; First posted 2018-08-06 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Progression From Impaired Fasting Glucose to Diabetes Mellitus
Keywords: Chinese; Diabetes Mellitus; Impaired fasting glucose; Incidence; Progression; Risk factors
MeSH Terms: conditions — Diabetes Mellitus; Disease Progression | interventions — Glucose Tolerance Test

STUDY DESIGN:
Intervention Model Description: Prospective and Cohort study (Compare different cohorts)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All recruited patients (Experimental): Blood taking procedure, oral glucose tolerance test and questionnaire will be included.
  Interventions: Diagnostic Test: Oral Glucose Tolerance Test; Diagnostic Test: HbA1c

INTERVENTIONS:
Diagnostic Test: Oral Glucose Tolerance Test — Patients will be invited to have oral glucose tolerance test. 2mL blood will be taken for analysis at 0 minute and 120 minutes.
Diagnostic Test: HbA1c — 2mL blood will be taken for analysis of HbA1c.

SUMMARY:
Impaired fasting glucose (IFG), a significant risk factor for diabetes mellitus (DM), is commonly encountered in the primary care setting and represents an important target for DM prevention. However, data on the long term risk of progression from IFG to DM among Chinese subjects and associated risk factors are currently lacking; appropriate DM prevention programme for this group cannot be yet established.

This is a prospective cohort study that aims to estimate the incidence of progression to diabetes mellitus (DM) among Chinese primary care patients with impaired fasting glucose (IFG) over a 3-year period and evaluate putative risk factors. A prospective cohort of around 700 non-diabetic Chinese adults who had IFG (i.e. fasting glucose level between 5.6 to 6.9mmol/L) and received baseline assessment between May 2013 and March 2015 at 3 public primary care clinics across Hong Kong will be invited for a 36-month-follow-up glycaemic status assessment (i.e. to repeat 75-gram oral glucose tolerance test (OGTT) and HbA1c test). The OGTT results will be used as the gold standard for the diagnosis of DM, normoglycaemia, IFG and impaired glucose tolerance (IGT) state. Demographics and lifestyle of the subjects including age, gender, occupation, education level, socio-economic status, smoking and drinking history, diet, exercise, work-sleep pattern, stress, quality of life and family history will be collected using standardized questionnaire. Participant's medical history and drug history will be retrieved from the Clinical Management System (CMS) of the Hospital Authority. Lipid profile, blood pressure, waist circumference and body mass index will also be assessed.

Logistic regression model will be performed to determine if these variables are associated with progression from IFG to DM. The primary outcome is the incidence of DM among the IFG study population. The secondary outcomes are the risks of developing DM among subjects with isolated IFG or combined IFG/IGT and determinants of progression to DM.

Knowledge on the natural history of isolated IFG or combined IFG/IGT among Hong Kong Chinese primary care patients and the significant modifiable associated risk factors for progression to DM will enable primary care researchers to design optimal management programme for diabetes prevention among these high risk patients.

DETAILED DESCRIPTION:
Impaired fasting glucose (IFG) represent an intermediate state of abnormal glucose regulation that exist between normal glucose homeostasis and diabetes mellitus (DM) and is a significant risk factor for DM and cardiovascular complications. IFG is defined by an elevated FG level between 6.1-6.9mmol/L according to the World Health Organization (WHO). The lower cutoff level for IFG was further lowered to 5.6mmol/L by the American Diabetes Association (ADA) in 2003 in order to maximize sensitivity and specificity for predicting DM over a 5-year period. In Hong Kong, IFG individuals can be more readily identified by primary care doctors than subjects with impaired glucose tolerance (IGT) or elevated HbA1c - the other 2 pre-diabetic categories - because fasting glucose (FG) test is recommended by the Hong Kong reference framework for diabetes care for adults in primary care setting for DM screening. Thus, this group of individuals should be targeted opportunistically for DM prevention.

On the other hand, IFG is a heterogeneous group with variable risk of progression to DM. Individuals with IFG may have concomitant IGT, elevated HbA1c or even DM. Thomas et al. found that around 20% of Hong Kong Chinese subjects with impaired glucose relation had concomitant IFG and IGT, whereas 49.5% had isolated IGT and 30.5% had isolated IFG. Ko et al. followed up 55 Chinese subjects with IFG for a median period of 1.12 year and showed that 8.4% progressed to DM annually as defined by fasting glucose criteria (FG ≥7.0mmol.L). Lee et al. followed up 238 Chinese women with persistent impaired glucose tolerance after gestational diabetes over a mean period of 52 months and found that 20% of the studied population developed diabetes mellitus based on OGTT criteria; the highest rate of progression to DM was noted among those women with concomitant postpartum impaired fasting glucose.

A recent cross-sectional study by Yu et al on 1,200 Chinese primary care patients with IFG demonstrated that 20% had DM confirmed by OGTT as the gold diagnostic standard, 14.3% had concomitant IGT, and 16.1% would regress back to normoglycaemia upon retest within 18 months. However, all of these local studies had short follow-up period and used different diagnostic tests for confirmation of DM; the long term risk of progression to DM among Chinese subjects with isolated IFG or combined IFG-IGT had not been fully evaluated.

Moreover, only few studies examined the risk factors for progression from IFG (+/- IGT) to DM among Asians or Chinese. Female gender, smoking, low physical activity, obesity as well as truncal obesity, high blood pressure, high triglyceridaemia and most importantly higher baseline FG level had all been reported to increase risk of progression from IFG to DM among Caucasians. In the only Asian study conducted in Japan, Toshihiro et al. found that stress in daily life, night duty and administrative position were risk factors of DM development among IFG subjects. To the best of our knowledge, no published data on the risk factors of progression from IFG to DM among Chinese is currently available. It was not certain that the risk factors identified among the Caucasians or Japanese were applicable to the Chinese. Although intensive lifestyle modifications targeting these risk factors had been reported to reduce progression from IFG to DM, their effects on Chinese subjects with IFG had not been evaluated.

Between May 2013 and March 2015, our team have already collected a prospective cohort of around 700 non-diabetic adults who have underwent both 75g OGTT and HbA1c tests as rigorous determination of their glycemic status. We aim to conduct a 3-year follow-up study to estimate the incidence of progression to DM among Hong Kong Chinese primary care patients with IFG with or without concomitant IGT using OGTT as the gold diagnostic standard as recommended by the Hong Kong Reference Framework. In addition, we aim to identify determinants, in particular the modifiable risk factors, for the progression from IFG to DM. These results will provide valuable information for designing optimal follow-up plan and diabetes prevention programme for local IFG patients, with the ultimate goal to reduce health care burden of DM on our society.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 18 year
2. Chinese ethnicity
3. Diagnosis of impaired fasting glucose (i.e. FG between 5.6-6.9mmol/L) +/- impaired glucose tolerance (i.e. 2-hour postprandial PG between 7.8-11.0mmol/L) confirmed by latest OGTT results within 60 months prior to recruitment

Exclusion Criteria:

* Confirmed diagnosis of DM or on hypoglycaemic treatment
* Women who are pregnant or breast-feeding at recruitment
* Patients taking glucocorticoid at recruitment
* Active and uncontrolled thyroid diseases (including subjects on thyroid replacement therapy or anti-thyroid drugs) or active endocrine diseases such as Cushing's syndrome or Acromegaly at recruitment
* Severe renal impairment i.e. eGFR ≤ 30 ml/min/1.73m2
* Clinically significant anaemia at recruitment
* History of blood donation or blood transfusion within 3 months prior to recruitment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 386 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-01-22 (Actual); Study Completion 2019-01-22 (Actual)

PRIMARY OUTCOMES:
Incidence of DM | At baseline
  the incidence of DM among Chinese primary care patients with impaired fasting glucose (including isolated IFG or combined IFG / IGT)

SECONDARY OUTCOMES:
Incidence of regression to normoglycaemia among the studied population | At baseline
Family history as risk factor associated with progression to DM | At baseline
  measured by questionnaire: ask if any direct relatives have the history of DM
Smoking habit as risk factor associated with progression to DM | At baseline
  measured by questionnaire: ask if participant is non-smoker, current smoker or ex-smoker
Drinking habit as risk factor associated with progression to DM | At baseline
  measured by questionnaire: ask if participant is non-drinker, social drinker, chronic drinker or ex-drinker
Stress level as risk factor associated with progression to DM | At baseline
  measured by questionnaire: Depression Anxiety Stress Scales (DASS) - 7 Stress Scales only
Stress level as risk factor associated with progression to DM | At baseline
  measured by questionnaire: Perceived Stress Scale (PSS-10)
Eating habit as risk factor associated with progression to DM | At baseline
  measured by diet questionnaire
Sleep quality as risk factor associated with progression to DM | At baseline
  measured by questionnaire Pittsburgh Sleep Quality Index (PSQI)
Exercises frequency as determinant of regression to normoglycaemia | At baseline
  measured by International Physical Activity Questionnaire (IPAQ) - short form
Diet as determinant of regression to normoglycaemia | At baseline
  measured by diet questionnaire
Sleep quality as determinants of regression to normoglycaemia | At baseline
  measured by Pittsburgh Sleep Quality Index (PSQI)
Waist circumferences as determinants of regression to normoglycaemia | At baseline
Prevalence of depression among subjects with IFG | At baseline
  measured by Patient Health Questionnaire (PHQ-2)
Health related Quality of Life of subjects with IFG | At baseline
  measured by questionnaire: SF12 Health Survey version 2
Capacity of the studied population to join intensive lifestyle intervention | At baseline
  by questionnaire: history of joining exercise classes or conducting diet control with dietitians

CONTACTS AND LOCATIONS:
Locations (3):
- Hong Kong (3):
  - Tsan Yuk Hospital RAMP Clinic, Hong Kong
  - Ap Lei Chau General Out-patient Clinic, Hong Kong
  - Lek Yuen General Out-patient Clinic, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] World Health Organization, Definition and diagnosis of diabetes mellitus and intermediate hyperglycaemia. 2006, World Health Organization: Geneva.
- [Background] Nathan DM, Davidson MB, DeFronzo RA, Heine RJ, Henry RR, Pratley R, Zinman B; American Diabetes Association. Impaired fasting glucose and impaired glucose tolerance: implications for care. Diabetes Care. 2007 Mar;30(3):753-9. doi: 10.2337/dc07-9920. No abstract available. PMID 17327355
- [Background] Genuth S, Alberti KG, Bennett P, Buse J, Defronzo R, Kahn R, Kitzmiller J, Knowler WC, Lebovitz H, Lernmark A, Nathan D, Palmer J, Rizza R, Saudek C, Shaw J, Steffes M, Stern M, Tuomilehto J, Zimmet P; Expert Committee on the Diagnosis and Classification of Diabetes Mellitus. Follow-up report on the diagnosis of diabetes mellitus. Diabetes Care. 2003 Nov;26(11):3160-7. doi: 10.2337/diacare.26.11.3160. No abstract available. PMID 14578255
- [Background] Task Force on Conceptual Model and Preventive Protocols, Hong Kong reference framework for diabetes care for adults in primary care settings. 2013: Hong Kong.
- [Background] Thomas GN, Schooling CM, McGhee SM, Ho SY, Cheung BM, Wat NM, Janus ED, Lam TH; Hong Kong Cardiovascular Risk Factor Prevalence Study Steering Committee. Identification of factors differentially associated with isolated impaired fasting glucose and isolated post-load impaired glucose tolerance: the Hong Kong Cardiovascular Risk Factor Study. Eur J Endocrinol. 2006 Oct;155(4):623-32. doi: 10.1530/eje.1.02250. PMID 16990663
- [Background] Ko GT, Chan JC, Cockram CS. Change of glycaemic status in Chinese subjects with impaired fasting glycaemia. Diabet Med. 2001 Sep;18(9):745-8. doi: 10.1046/j.0742-3071.2001.00572.x. PMID 11606173
- [Background] Lee KF, Mak MW, Lau KO, Chung H. Risk of development of diabetes mellitus in Chinese women with persistently impaired glucose tolerance after gestational diabetes. Hong Kong Med J. 2011 Jun;17(3):195-201. PMID 21636867
- [Background] Yu EY, Wong CK, Ho SY, Wong SY, Lam CL. Can HbA1c replace OGTT for the diagnosis of diabetes mellitus among Chinese patients with impaired fasting glucose? Fam Pract. 2015 Dec;32(6):631-8. doi: 10.1093/fampra/cmv077. Epub 2015 Oct 14. PMID 26467644
- [Background] Rasmussen SS, Glumer C, Sandbaek A, Lauritzen T, Borch-Johnsen K. Determinants of progression from impaired fasting glucose and impaired glucose tolerance to diabetes in a high-risk screened population: 3 year follow-up in the ADDITION study, Denmark. Diabetologia. 2008 Feb;51(2):249-57. doi: 10.1007/s00125-007-0893-8. Epub 2007 Dec 5. PMID 18060659
- [Background] Leiva E, Mujica V, Orrego R, Wehinger S, Soto A, Icaza G, Vasquez M, Diaz L, Andrews M, Arredondo M. Subjects with impaired fasting glucose: evolution in a period of 6 years. J Diabetes Res. 2014;2014:710370. doi: 10.1155/2014/710370. Epub 2014 Aug 20. PMID 25215305
- [Background] Nichols GA, Hillier TA, Brown JB. Progression from newly acquired impaired fasting glusose to type 2 diabetes. Diabetes Care. 2007 Feb;30(2):228-33. doi: 10.2337/dc06-1392. PMID 17259486
- [Background] Sharifi F, Jaberi Y, Mirzamohammadi F, Mirzamohammadi H, Mousavinasab N. Determinants of developing diabetes mellitus and vascular complications in patients with impaired fasting glucose. Indian J Endocrinol Metab. 2013 Sep;17(5):899-905. doi: 10.4103/2230-8210.117240. PMID 24083174
- [Background] Toshihiro M, Saito K, Takikawa S, Takebe N, Onoda T, Satoh J. Psychosocial factors are independent risk factors for the development of Type 2 diabetes in Japanese workers with impaired fasting glucose and/or impaired glucose tolerance. Diabet Med. 2008 Oct;25(10):1211-7. doi: 10.1111/j.1464-5491.2008.02566.x. PMID 19046200
- [Background] Knowler WC, Barrett-Connor E, Fowler SE, Hamman RF, Lachin JM, Walker EA, Nathan DM; Diabetes Prevention Program Research Group. Reduction in the incidence of type 2 diabetes with lifestyle intervention or metformin. N Engl J Med. 2002 Feb 7;346(6):393-403. doi: 10.1056/NEJMoa012512. PMID 11832527